CLINICAL TRIAL: NCT02463266
Title: Evaluation of the PACE/PACENET BHL Clinical Program
Acronym: SUSTAINIV
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Magellan Health Services (Other)
Responsible Party: Principal Investigator, Mary Beth Gibbons, Ph.D., Professor of Psychiatry, Director of Center for Psychotherapy Research, Department of Psychiatry University of Pennsylvania, University of Pennsylvania
Other Study IDs: 819712
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anxiety; Pain, Chronic
Keywords: Primary Care; Elderly; Depression
MeSH Terms: conditions — Depression; Anxiety Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- SUSTAIN Monitoring and Care Management: SUSTAIN program participants who complete an initial clinical assessment and, if indicated, agree to follow-up services including Monitoring and/or Care Management.
  Interventions: Behavioral: SUSTAIN Monitoring and Care Management

INTERVENTIONS:
Behavioral: SUSTAIN Monitoring and Care Management — Program participants are offered clinical services based on symptom severity and clinical need. Follow-up Monitoring consists of up to 4 brief, structured assessments following the baseline clinical assessment. These follow-up contacts are conducted over the telephone by the HT/BHP and take place during the initial 12 weeks of pharmaceutical treatment. These brief interviews monitor symptoms, adherence, side effects, and response to treatment. Care Management incorporates the use of a BHP who has expertise in mental health assessment and is well versed in the delivery of algorithm-based management strategies. The BHP monitors and encourages patient acceptance and adherence to treatment recommendations through support, education, and motivational engagement.

SUMMARY:
The SUpporting Seniors Receiving Treatment And INtervention (SUSTAIN) program is a telephone-based clinical service designed to help identify and manage behavioral health issues among PACE/PACENET enrollees. The purpose of the current project is to a) explore moderators of treatment response among beneficiaries in the SUSTAIN Clinical Program and b) to evaluate the sustained clinical effects of the program.

DETAILED DESCRIPTION:
The SUpporting Seniors Receiving Treatment And INtervention (SUSTAIN) program is an evidence-based clinical service administered via telephone and designed to help identify and manage behavioral health issues among enrollees of the Commonwealth of Pennsylvania Department of Aging's Pharmaceutical Assistance Contract for the Elderly (PACE) and the PACE Needs Enhancement Tier (PACENET) Program who have been newly prescribed psychotropic medications. The SUSTAIN program has adapted the existing software and staffing model from Penn's Behavioral Health Laboratory (BHL), which has been used to integrate Mental Health (MH) care within primary care in other health systems, including the VA where it was originally developed. The SUSTAIN program is a novel and flexible clinical service that addresses some of the barriers that hinder treatment outcomes for MH problems. Given the fact that the SUSTAIN program provides assessment, monitoring, early intervention, disease management, and referral management over the telephone, the program can be tailored to each individual's specific needs. The SUSTAIN program also overcomes logistical barriers such as the necessity of frequent face-to-face contact in specialty programs, and thus can enhance existing specialty care programs by reducing wait times and "no-show" rates. As a result, the SUSTAIN program has the potential to result in higher patient satisfaction, improved health, and, accordingly, greater independent functioning.

The SUSTAIN program assesses individuals with behavioral health issues and offers a subset of these individuals ongoing follow-up services based on clinical need and symptom severity. Follow-up service options include Monitoring and Care Management. Monitoring consists of up to 4 brief (5-10 minutes), structured assessments following the baseline assessment. These follow-up contacts are conducted over the telephone by the Heath Technician (HT) or Behavioral Health Provider (BHP) and take place during the initial 12 weeks of pharmaceutical treatment. These brief interviews monitor symptoms, adherence, side effects, and response to treatment. Care Management is algorithm-driven care for conditions such as depression, panic disorder, generalized anxiety disorder, and chronic pain, and is delivered by a BHP as an adjunct to primary care. The BHP monitors and encourages patient acceptance and adherence to treatment recommendations through support, education, and motivational engagement.

The investigators will evaluate the extent to which SUSTAIN is related to program participants' outcomes. The evaluation of the program relies on 2 sources of data: 1) a retrospective chart review of data collected as part of the clinical program, which includes data from the baseline and follow-up clinical interviews, and 2) data collected during a one-time 6 Month Outcome Research Evaluation interview completed with SUSTAIN program participants who provide verbal consent. The retrospective chart review will evaluate the clinical data from 5500 PACE/PACENET enrollees who participate in the PACE/PACENET SUSTAIN Clinical Program (which includes both Monitoring and Care Management). The 6 Month Outcome Research Evaluation will evaluate long term outcomes among a subset of participants.

Clinical Program Procedures:

Referred PACE/PACENET enrollees are contacted to complete an initial baseline clinical interview. Following the baseline interview, enrollees are offered several different services, depending on clinical need: Referral Management, Care Management, or Monitoring. Enrollee participation in the program occurs over the span of up to six months, with the number of calls based upon the follow-up service.

Study Procedures:

A. Retrospective Chart Review Procedures:

The retrospective chart review of the clinical data (i.e., data collected at baseline and during Monitoring and Care Management visits) will be conducted and saved as a separate research database. The research database will be de-identified (but include coded data) and kept in a separate password protected file.

B. 6 Month Outcome Research Evaluation Procedures:

PACE/PACENET enrollees who participate in the SUSTAIN Clinical Program will be asked to provide verbal HIPAA authorization and consent for participation in the 6 Month Outcome Research Evaluation at the end of the acute phase of clinical care, usually at three months. Enrollees providing verbal consent to participate in the 6 Month Outcome Research Evaluations will be called again at 6 months following the date of the initial clinical interview. At the 6 Month Outcome Research call, assessments will be conducted that mirror the SUSTAIN Clinical Program baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 and older, males and females.
2. Participating in the SUSTAIN Clinical Program
3. For the 6 Month Outcome Research Evaluation, in addition to meeting criteria 1 and 2, willing to provide verbal informed consent to participate in the 6 Month Outcome Research Evaluation at the end of the acute phase of clinical care, usually at three months.

Exclusion Criteria:

* Not meeting the inclusion criteria listed above.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: PACE/PACENET beneficiaries who are participating in the PACE/PACENET SUSTAIN Clinical Program.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Veterans Rand - 12 Item Health Survey (VR-12) | 6 months
  A measure of physical and mental health functioning

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 item Scale (PHQ-9) | 6 months
  A measure of depression severity
Generalized Anxiety Disorder - 7 item Scale (GAD-7) | 6 months
  A measure of anxiety severity

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Gibbons, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Department of Psychiatry (Center for Psychotherapy Research), University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maust DT, Chen SH, Benson A, Mavandadi S, Streim JE, DiFilippo S, Snedden TM, Oslin DW. Older adults recently started on psychotropic medication: where are the symptoms? Int J Geriatr Psychiatry. 2015 Jun;30(6):580-6. doi: 10.1002/gps.4187. Epub 2014 Aug 12. PMID 25116369
- [Background] Maust DT, Mavandadi S, Benson A, Streim JE, Difilippo S, Snedden T, Weber AL, Oslin DW. Telephone-based care management for older adults initiated on psychotropic medication. Int J Geriatr Psychiatry. 2013 Apr;28(4):410-6. doi: 10.1002/gps.3839. Epub 2012 Jun 7. PMID 22678956
- [Background] Oslin DW, Ross J, Sayers S, Murphy J, Kane V, Katz IR. Screening, assessment, and management of depression in VA primary care clinics. The Behavioral Health Laboratory. J Gen Intern Med. 2006 Jan;21(1):46-50. doi: 10.1111/j.1525-1497.2005.0267.x. PMID 16423122
- [Background] Maust DT, Mavandadi S, Eakin A, Streim JE, Difillipo S, Snedden T, Oslin DW. Telephone-based behavioral health assessment for older adults starting a new psychiatric medication. Am J Geriatr Psychiatry. 2011 Oct;19(10):851-8. doi: 10.1097/JGP.0b013e318202c1dc. PMID 21946801
- [Background] Mavandadi S, Benson A, DiFilippo S, Streim JE, Oslin D. A Telephone-Based Program to Provide Symptom Monitoring Alone vs Symptom Monitoring Plus Care Management for Late-Life Depression and Anxiety: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1211-8. doi: 10.1001/jamapsychiatry.2015.2157. PMID 26558530
- [Background] Gerlach LB, Mavandadi S, Maust DT, Streim JE, Oslin DW. Improving Access to Collaborative Behavioral Health Care for Rural-Dwelling Older Adults. Psychiatr Serv. 2018 Jan 1;69(1):117-120. doi: 10.1176/appi.ps.201700026. Epub 2017 Oct 2. PMID 28967325
- [Background] Gerlach LB, Maust DT, Leong SH, Mavandadi S, Oslin DW. Factors Associated With Long-term Benzodiazepine Use Among Older Adults. JAMA Intern Med. 2018 Nov 1;178(11):1560-1562. doi: 10.1001/jamainternmed.2018.2413. PMID 30208384